CLINICAL TRIAL: NCT00205725
Title: Glucose Regulation During Ziprasidone Treatment
Brief Title: Pfizer/IVGTT/Ziprasidone/Olanzapine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pfizer IVGTT/941273
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia; Type 2 Diabetes Mellitus
Keywords: Schizophrenia; BMI; T2DM
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus, Type 2 | interventions — ziprasidone; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ziprasidone, Olanzapine

SUMMARY:
Abnormalities in peripheral glucose regulation and type 2 diabetes can occur more commonly in individuals with schizophrenia than in healthy subjects or in other psychiatric conditions. Antipsychotic treatment may contribute significantly to abnormalities in glucose regulation. Hyperglycemia can contribute to long-term cardiovascular disease risk that may already be increased in patients with schizophrenia due to higher rates of smoking, sedentary life style, obesity and under-treated hypertension and dyslipidemia. This project will characterize the effects on glucose control of the two most commonly prescribed newer antipsychotic medications, ziprasidone and olanzapine, in patients with schizophrenia.

DETAILED DESCRIPTION:
This proposal aims to use a well-characterized procedure, the modified Frequently Sampled Intravenous Glucose Tolerance Test (FSIGTT), to characterize the glucoregulatory effects of the two most commonly prescribed atypical antipsychotic medications, ziprasidone and olanzapine, in comparison to the conventional antipsychotic haloperidol. Abnormalities in peripheral glucose regulation and type 2 diabetes can occur more commonly in individuals with schizophrenia than in healthy subjects or in other psychiatric conditions. While abnormalities in glucose regulation were first reported in schizophrenia prior to the introduction of antipsychotic medications, antipsychotic treatment may contribute significantly to abnormalities in glucose regulation.

Recently, the adverse effect of antipsychotic medications on systemic glucose regulation has received increased attention as investigators noted prominent adverse glucoregulatory effects associated with certain newer antipsychotic medications. Abnormal glucose regulation and new-onset type 2 diabetes have been reported during clozapine and olanzapine treatment. Complicating the study of antipsychotic-induced changes in glucose regulation, increased adiposity can decrease insulin sensitivity, and antipsychotics can increase adiposity and body mass index (BMI). However, abnormal glucose regulation and type 2 diabetes can occur during clozapine treatment in the absence of weight gain, suggesting that changes in glucose regulation can occur independent of drug-induced increases in BMI. Consistent with this, our preliminary studies indicate that important effects of clozapine and olanzapine on glucose regulation are not accounted for by differences in BMI. This proposal will compare the effects of olanzapine, ziprasidone and haloperidol on well-defined measures of glucose regulation.

This proposal specifically hypothesizes that olanzapine treatment will be associated with decreases in insulin sensitivity (SI), without effects on insulin secretion. Treatment-related effects on glucose effectiveness (SG) will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients: meets DSM-IV criteria for schizophrenia, any type, or schizoaffective disorder;
* aged 18 to 60 years;
* able to give informed consent;
* no medication changes for 2 weeks prior to and during the period of study;
* Patients: currently taking an antipsychotic.

Exclusion Criteria:

* Controls: Axis I psychiatric disorder criteria met except for substance use disorders as below;
* meets DSM-IV criteria for the diagnoses of substance abuse or dependence within the past six months;
* involuntary legal status (as per Missouri law);
* the presence of any serious medical disorder that may (as confirmed by peer-reviewed literature) confound the assessment of symptoms, relevant biologic measures or diagnosis;
* the following conditions are currently identified:

  * insulin- or non-insulin-dependent diabetes mellitus;
  * any intra-abdominal or intrathoracic surgery or limb amputation within the prior 6 months;
  * any diagnosed cardiac condition causing documented hemodynamic compromise;
  * any diagnosed respiratory condition causing documented or clinically recognized hypoxia;
  * pregnancy or high dose estrogens, fever, narcotic therapy, acute sedative hypnotic withdrawal, corticosteroid or spironolactone therapy, dehydration, epilepsy, endocrine disease, high-dose benzodiazepine therapy (> 25 mg/day of diazepam), or any medical condition known to interfere with glucose utilization;
* meets DSM-IV criteria for Mental Retardation (mild or worse).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2000-11; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Effects of olanzapine/ziprasidone/haloperidol on glucose regulation

SECONDARY OUTCOMES:
Explore treatment-related effects on glucose effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: John W. Newcomer, M.D., Principal Investigator — Washington University School of Medicine and Florida Atlantic University
Locations (1):
- Washington University School of Medicine, Psychiatry Dept., St Louis, Missouri, United States

REFERENCES:
- [Result] Haupt DW, Fahnestock PA, Flavin KA, Schweiger JA, Stevens A, Hessler MJ, Maeda J, Yingling M, Newcomer JW. Adiposity and insulin sensitivity derived from intravenous glucose tolerance tests in antipsychotic-treated patients. Neuropsychopharmacology. 2007 Dec;32(12):2561-9. doi: 10.1038/sj.npp.1301392. Epub 2007 Mar 21. PMID 17375138
- [Result] Haupt DW, Luber A, Maeda J, Melson AK, Schweiger JA, Newcomer JW. Plasma leptin and adiposity during antipsychotic treatment of schizophrenia. Neuropsychopharmacology. 2005 Jan;30(1):184-91. doi: 10.1038/sj.npp.1300563. PMID 15367925